CLINICAL TRIAL: NCT05300386
Title: Using Wearable Devices to Investigate the Basic Physical Conditions of Patients With Sleep Problems and the Physical Effects During Sleep on Patients Who Use the Central Nervous Medications for Sleep Problems
Brief Title: Wearable Devices to Assess Effects of Central Nervous Medications on Physical Conditions in Patients With Sleep Problems
Status: Completed | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Tien-Yu Chen, Visiting Physician, Tri-Service General Hospital
Other Study IDs: 2-107-05-046
Record Dates: First submitted 2022-02-26; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Anxiety Disorders; Sleep Apnea
Keywords: anxiety; sleep apnea
MeSH Terms: conditions — Anxiety Disorders; Sleep Apnea Syndromes | interventions — Escitalopram

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- generalized anxiety with oxygen desaturation index less than 5: we enrolled patients with generalized anxiety with oxygen desaturation index of less than 5 and examed the basic physical conditions and the effectiveness of antidepressant treatment.
  Interventions: Drug: Escitalopram
- generalized anxiety with oxygen desaturation index more than 5: we enrolled patients with generalized anxiety with oxygen desaturation index of more than 5 and examed the basic physical conditions and the effectiveness of antidepressant treatment.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — We use Escitalopram 5~10 mg for two groups to observe the impact of sleep apnea on the treatment of generalized anxiety disorder

SUMMARY:
Generalized anxiety disorder (GAD) and obstructive sleep apnea (OSA) are two common diseases and share similar symptoms such as anxiety, poor attention, and poor sleep quality. However, the evidence toward the association between GAD and OSA is limited. The current study aims to use wearable devices to detect comorbid OSA in newly diagnosed patients with GAD and observe the treatment response and difference in automatic nervous function in GAD and GAD/OSA groups.

DETAILED DESCRIPTION:
Background: The symptoms of a generalized anxiety disorder (GAD) included excessive anxiety, restlessness, fatigue, poor concentration, irritability, and poor sleep quality. GAD is frequently combined with depressive disorder and autonomic dysfunction and is one of the most prevalent psychiatric disorders in a psychiatric clinic. However, many of the symptoms of GAD are like the symptoms of obstructive sleep apnea (OSA), such as daytime fatigue, poor attention, and poor sleep quality. In addition, patients with OSA are easily comorbid with symptoms of anxiety and depression in retrospective studies. Nevertheless, there is limited data present on the comorbid of OSA in newly diagnosed patients with GAD. It is important to realize the comorbidities between OSA and GAD. Many of the benzodiazepines for GAD during sleep may worsen the severity of sleep apnea. Therefore, realizing the relationship between GAD and OSA is important for clinicians.

Question/Hypothesis: We hypothesize that patients with newly diagnosed GAD have a high ratio of OSA comorbidity and those with both GAD and OSA have worse severity of anxiety symptoms and heart rate variability.

Specific Aims: Current study aims to investigate 1) the prevalence of OSA in newly diagnosed patients with GAD; 2) the difference of heart rate variability and baseline characteristics between newly diagnosed patients with GAD and GAD with OSA; 3) the difference of antidepressant treatment response between newly diagnosed patients with GAD and GAD with OSA.

Experimental design: This study aims to enroll 80 participants with GAD, 40 patients with newly diagnosed GAD and 40 newly diagnosed GAD comorbid with OSA by using a home sleep apnea test and used validated cloud-computing sleep apnea screening system. In addition, we would investigate the difference between baseline characteristics and heart rate variability among healthy participants, GAD, and GAD comorbid OSA. In addition, we also evaluate the difference in antidepressant treatment effect on GAD patients with and without OSA on week 2, week 4, and week 12.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis as drug-naïve GAD with an unexpected diagnosis of OSA
* Go to bed between 8:30 pm to midnight
* Have a BMI between 18-34
* Agree to sign an informed consent and use wearable devices to detect sleep

Exclusion Criteria:

* Pregnancy and pacemaker implantation
* Shift workers or travel to 3 different timelines 7 days before study entry day
* Diabetes, cancer, neuropathy, any cardiovascular diseases that affect HRV
* Alcohol, illegal drugs, tobacco use
* Currently use medications that affect the HRV (e.g., antipsychotics, anticholinergics, antidepressants, and anticonvulsants)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Taiwanese
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2021-05-29 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change of the severity of anxiety measured by Beck Anxiety Inventory (BAI) across three points of the study | Assessed at the second, fourth, and twelfth weeks of the study
  The Beck Anxiety Inventory (BAI) is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in adolescents and adults ages 17 and older. The questions used in this measure ask about common symptoms of anxiety that the subject has had during the past week (including the day you take it) (such as numbness and tingling, sweating not due to heat, and fear of the worst happening). The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms.
  The standardized cutoffs are:
  * 0-7: Minimal
  * 8-15: Mild
  * 16-25: Moderate
  * 26-63: Severe
Change of the severity of depression measured by Beck Depression Inventory (BDI) across three points of the study | Assessed at the second, fourth, and twelfth weeks of the study
  The Beck Depression Inventory (BDI) is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. The BDI is designed for individuals aged 13 and over, and is composed of items relating to symptoms of depression such as hopelessness and irritability, cognitions such as guilt or feelings of being punished, as well as physical symptoms such as fatigue, weight loss, and lack of interest in sex. The BDI contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms.
  The standardized cutoffs are:
  * 0-13: minimal depression
  * 14-19: mild depression
  * 20-28: moderate depression
  * 29-63: severe depression.
Change of the severity of daytime sleepiness measured by Epworth Sleepiness Scale (ESS) across three points of the study | Assessed at the second, fourth, and twelfth weeks of the study
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
  In general ESS scores can be interpreted as follows:
  * 0-5 Lower Normal Daytime Sleepiness
  * 6-10 Higher Normal Daytime Sleepiness
  * 11-12 Mild Excessive Daytime Sleepiness
  * 13-15 Moderate Excessive Daytime Sleepiness
  * 16-24 Severe Excessive Daytime Sleepiness
Change of sleep quality measured by Pittsburgh Sleep Quality Index (PSQI) across three points of the study | Assessed at the second, fourth, and twelfth weeks of the study
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. The PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. A final score >5 be considered as a significant sleep disturbance.
Change of autonomic nervous system functioning measured by Heart rate variability (HRV) across three points of the study | Assessed at the second, fourth, and twelfth weeks of the study
  Heart rate variability (HRV) consists of changes in the time intervals between consecutive heartbeats called interbeat intervals (IBIs). HRV indexes neurocardiac function and is generated by heart-brain interactions and dynamic non-linear autonomic nervous system processes. HRV reflects regulation of autonomic balance, blood pressure (BP), gas exchange, gut, heart, and vascular tone, which refers to the diameter of the blood vessels that regulate BP, and possibly facial muscles. HRV can be analyzed through time-domain, frequency-domain, and non-linear metrics. Time-domain indices quantify the amount of HRV observed during monitoring periods that may range from ~2 min to 24 h. Frequency-domain values calculate the absolute or relative amount of signal energy within component bands. Non-linear measurements quantify the unpredictability and complexity of a series of IBIs.

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Yu Chen, MD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Neihu, Taiwan